CLINICAL TRIAL: NCT02489604
Title: Peptide Receptor Radionuclide Therapy (PRRT) with Radiolabelled Somatostatin Analogue 177Lu-DOTATATE in Advanced Gastro-entero Pancreatic Neuroendocrine Tumors, 18F-2-fluoro-2-deoxy-D-glucose (FDG)-PET Negative Patients: a Prospective Phase II Randomized Study
Brief Title: Peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-DOTATATE in Advanced Gastro-entero Pancreatic Neuroendocrine Tumors
Acronym: LUNET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment target not reached
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.11
Record Dates: First submitted 2015-06-16; First posted 2015-07-03 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 177Lu-DOTATATE 25.9 GBq activity (Experimental): 177Lu-DOTATATE 25.9 GBq activity. Total activity of 25.9 GBq 100 mCi for 7 cycles every 6 ± 2 weeks (700 mCi)
  Interventions: Drug: 177Lu-DOTATATE 25.9 GBq activity
- 177Lu-DOTATATE 18.5 GBq activity (Experimental): 177Lu-DOTATATE 18.5 GBq activity. Total activity of 18.5 GBq 100 mCi for 5 cycles, every 6 ± 2 weeks (500 mCi)
  Interventions: Drug: 177Lu-DOTATATE 18.5 GBq activity

INTERVENTIONS:
Drug: 177Lu-DOTATATE 25.9 GBq activity — 177Lu-DOTATATE will be administered in a 30 minutes infusion. Total activity of 25.9 GBq 100 mCi for 7 cycles every 6 ± 2 weeks (700 mCi)
  Other Names: 177Lu-DOTATATE
  Arms: 177Lu-DOTATATE 25.9 GBq activity
Drug: 177Lu-DOTATATE 18.5 GBq activity — 177Lu-DOTATATE will be administered in a 30 minutes infusion Total activity of 18.5 GBq 100 mCi for 5 cycles , every 6 ± 2 weeks (500 mCi)
  Other Names: 177Lu-DOTATATE
  Arms: 177Lu-DOTATATE 18.5 GBq activity

SUMMARY:
This is a randomized phase II non-comparative study. Patients with gastroenteropancreatic Neuroendocrine tumour (GEP-NET) G1-G2 with progressive disease, SSR positive and FDG negative will be enrolled in the study and will be randomly assigned to 2 different dosages (total activity of 25.9 GBq and total activity of 18.5 GBq).

DETAILED DESCRIPTION:
This is a randomized phase II non-comparative study. Patients with GEP-NET G1-G2 with progressive disease, somatostatin receptor (SSR) positive and FDG negative will be enrolled in the study and will be randomly assigned to 2 different dosages (total activity of 25.9 GBq and total activity of 18.5 GBq). The two levels of dosages are:

1. Total activity of 25.9 GBq 100 mCi for 7 cycles at 6 ± 2 weeks (700 mCi)
2. Total activity of 18.5 GBq 100 mCi for 5 cycles at 6 ± 2 weeks (500 mCi) The randomized study design allows for two active treatments to be evaluated in a comparable patient population. The estimates of primary objectives can be evaluated for each regimen separately by a Bryant and Day design. While the sample size is not powered for statistical test of a specific hypothesis for comparison between groups, this study design allows the unbiased collection of activity and safety in these two regimens in the same population, which will be useful for planning future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmation of GEP -NETand Ki 67 index <= 20%.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1.criteria)
* Advanced GEP-NET are eligible; patients must have progressive disease based on RECIST 1.1. criteria
* Diagnostic OctreoScan and/or PET/CT 68Ga-peptide images demonstrate a significant uptake in the tumour
* FDG PET negative (SUV less than 2.5)
* Concomitant somatostatin analogs assumption is allowed
* Life expectancy greater than 6 months.
* ECOG performance status <2
* Adequate haematological, liver and renal function: haemoglobin >= 9 g/dL, absolute neutrophil count (ANC) >= 1.5 x 109 /L, platelets >= 100 x 109 /L, bilirubin ≤1.5 X upper normal limit (UNL) , Alanine transaminase (ALT) <2.5 X UNL (< 5 X UNL in presence of liver metastases), creatinine < 2 mg/dL.
* If female of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug. Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Ki 67 index > 20 %
* FDG PET positive at least in one documented lesion with a SUV more than 2.5
* Patients treated with chemotherapy and therapeutic radiotherapy within 4 weeks and treated within 2 weeks with palliative radiotherapy, hormonal or biological therapy).
* Patients treated with previous radiometabolic therapy with an adsorbed dose to the kidney more than 25 Gy and 1,5 Gy for the bone marrow.
* All acute toxic effects of any prior therapy (including surgery radiation therapy, chemotherapy) must have resolved to a grade <= 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE)
* Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-12; Primary Completion 2024-01 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) | up to 7 years
  the complete response rate plus the partial response rate plus the rate of patients with stable disease for at least 12 months from therapy start on patient population randomly assigned to two different scheme of therapy
Acute toxicity evaluated according to version 4.0 CTCAE | The evaluation of the acute toxicity starts from the 1st treatment until 30 days after the last treatment cycle, up to 60 wks for each patient
  The co-primary objective is the acute toxicity evaluated according to version 4.0 CTCAE

SECONDARY OUTCOMES:
Progression free survival | up to 7 years
  the time from the start treatment date to the date of first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
Overall survival | up to 7 years
  Overall survival is defined as the time from the therapy start to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.
Late toxicity evaluated according to version 4.0 CTCAE | up to 7 years
  late toxicity will be evaluated during the whole study period according to version 4.0 CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Sansovini, MD, Principal Investigator — IRST IRCCS
Locations (1):
- Irst Irccs, Meldola, FC, Italy